CLINICAL TRIAL: NCT02661165
Title: Exploratory Study: How Does the Spirituality of a Group of British People With Type 2 Diabetes Impact Their Coping and Self-management of Their Condition?
Brief Title: How Does the Spirituality of Patients With Type 2 Diabetes Influence Their Self-management?
Status: Completed | Type: Observational
Sponsor: Natasha Duke (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor-Investigator, Natasha Duke, Doctoral Student, University of Southampton
Organization: University of Southampton (Other)
Other Study IDs: USouthampton
Record Dates: First submitted 2015-12-17; First posted 2016-01-22 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This exploratory study is researching how the spirituality of a group of British patients with type 2 diabetes (T2D), impacts their approach to the self-management of their condition.

Bio-statistical markers will be taken from consenting participants' Clinic database records. Qualitative interviews will be conducted with participants, and the results analysed and interpreted, alongside their bio-statistical markers.

Results will be presented in healthcare peer reviewed journals and conferences, to inform clinicians how patients' self-management of their T2D is influenced by their spirituality.

DETAILED DESCRIPTION:
Patients will be recruited from diabetes clinics.

The bio-statistical markers will be: include their living situation (living alone or with family/partner); date of T2D diagnosis; current age; glycated haemoglobin (hba1c) blood test; body mass index and current pharmacological therapy. This data will be collected from the Diabetes Clinic to contextualize the qualitative data. These measurements will reveal how well a participant is managing their T2D.

The Biographic Narrative Interpretive Method (BNIM) will involve interviews with eight participants. Each participant will have at least 2 and possibly 3 interviews at a location of their choice. The data will undergo thematic analysis, which will be interpreted.

The results will be used to encourage clinicians to consider the spirituality of people with T2D when planning their care, thus giving holistic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Speak English
* Have had T2D at least 6 months.
* Have read the Participant Information Sheet, explaining this study is regarding T2D, spirituality, coping and self-management.
* Gives consent to access their diabetes details that are stored on a Clinic database.
* Gives consent to recorded interviews.

Exclusion Criteria:

* Not speak English.
* Have had T2D less than 6 months.
* Have read the Participant Information Sheet, and decided they are not comfortable talking about their T2D, or spirituality, or coping or their self-management.
* Not consenting to data collection from Clinic records.
* Clinic records have not been kept (e.g. is a new patient to their family doctor).
* Consent is withdrawn from the study (which could be any stage).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with T2D from a community or primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-06; Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
The self-management Interviews to identify if and how patients' spirituality influences their diet and exercise. | 58 months
  An exploratory study using qualitative data only to identify if and how patients' spirituality influences their diet and exercise, both of which are key to good diabetes control, and the prevention of diabetic complications in the long term. (No quantitative data will be collected, and as such no outcome measures will be collected).
  Interviews will utilize the biographical narrative interpretive method to reveal how beliefs may influence diet and exercise. Each interview may last up to 3 hours. Each participant will be interviewed up to 3 times (approximately 9 hours of interviewing per participant). Interviews will be transcribed verbatim. Themes will be generated, coded and interpreted. Results will be the researchers interpretive analysis of the qualitative data generated, and the themes that emerge.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Duke, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT02661165/Prot_ICF_000.pdf